CLINICAL TRIAL: NCT05061004
Title: Cephea Early Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10354
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment of symptomatic patients with mitral valve disease (including mitral regurgitation, mitral stenosis and mixed mitral valve disease) with the Cephea Mitral Valve System
  Interventions: Device: Cephea Mitral Valve System

INTERVENTIONS:
Device: Cephea Mitral Valve System — Transcatheter mitral valve replacement

SUMMARY:
The objective of this study is to evaluate the preliminary safety and effectiveness of the Cephea Mitral Valve System for the treatment of symptomatic patients with mitral valve disease (including mitral regurgitation, mitral stenosis and mixed mitral valve disease) in whom transcatheter therapy is deemed more appropriate than open heart surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* Mitral valve disease resulting in mitral regurgitation (MR ≥ Grade III) and/or severe mitral valve stenosis (mitral valve area ≤ 1.5cm²) per American Society of Echocardiography criteria.
* LVEF ≥ 30%
* In the judgement of the Site Heart Team, transcatheter therapy is deemed more appropriate than open heart surgery.

Key Exclusion Criteria:

* Prior surgical or interventional treatment that interferes with the Cephea valve delivery or function.
* Need for emergent or urgent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 30 days post implant
  Freedom from all-cause mortality, which will be assessed at 30 days post implant.
Primary Effectiveness Endpoint | 30 days post implant
  Proportion of subjects with reduction of MR to ≤ Grade I, will be assessed at 30 days post implant.

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott Structural Heart
Locations (22):
- United States (20):
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Davis Medical Center, Sacramento, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - University of Michigan - Davis Medical Center, Ann Arbor, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Atrium Health - Carolinas Medical Center, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - Ascension Saint Thomas, Nashville, Tennessee
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Houston Methodist, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
- Canada (2):
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Institut de Cardiologie de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No